CLINICAL TRIAL: NCT05532085
Title: Assessment of Pain During Voluntary Termination of Pregnancy Following Consideration of Predictive Factors of Pain, With and Without an Established Analgesic Protocol.
Brief Title: Assessment of Pain During an Abortion With Knowledge of the Predictive Factors of Pain.
Status: Completed | Type: Observational
Sponsor: Olivier CHASSANY (Other)
Responsible Party: Sponsor-Investigator, Olivier CHASSANY, Professor, University Paris 7 - Denis Diderot
Organization: University Paris 7 - Denis Diderot (Other)
Other Study IDs: ED-IVG
Record Dates: First submitted 2022-05-27; First posted 2022-09-08 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Induced Abortion; Medical Abortion; Surgical Abortion; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group: Medical abortion without analgesic protocol: All women over the age of 15, benefiting from a medical abortion between June and October 2020, including oral French.
  Interventions: Other: Evaluation of pain during voluntary termination of pregnancy with medication following consideration of predictive factors of pain without an established analgesic protocol
- Group: Medical abortion with analgesic protocol: All women over the age of 15, benefiting from a medical abortion between October 2020 and February 2021, including spoken French.
  Interventions: Other: Evaluation of pain during a voluntary medical termination of pregnancy following consideration of predictive factors of pain with an established analgesic protocol
- Group: Abortion by aspiration under local anesthesia without analgesic protocol: All women over the age of 15, benefiting from an abortion by aspiration under local anesthesia between June and October 2020, including oral French.
  Interventions: Other: Assessment of pain during voluntary termination of pregnancy by aspiration under local anesthesia following consideration of predictive factors of pain without an established analgesic protocol
- Group: Abortion by aspiration under local anesthesia with analgesic protocol: All women over the age of 15, benefiting from an abortion by aspiration under local anesthesia between October 2020 and February 2021, including oral French.
  Interventions: Other: Assessment of pain during voluntary termination of pregnancy by aspiration under local anesthesia following consideration of predictive factors of pain with established analgesic protocol

INTERVENTIONS:
Other: Evaluation of pain during voluntary termination of pregnancy with medication following consideration of predictive factors of pain without an established analgesic protocol — Evaluation of the pain felt by women having an abortion by aspiration under local anes!thesia.
  The intensity of the pain of patients during an abortion by aspiration under local anesthesia will be quantified by a Visual Analogue Scale (VAS) at the time of the abortion and in the following 4 days.
  Groups: Group: Medical abortion without analgesic protocol
Other: Evaluation of pain during a voluntary medical termination of pregnancy following consideration of predictive factors of pain with an established analgesic protocol — Evaluation of the pain felt by women having a medical abortion following the application of an analgesic protocol indexed on the predictive factors of pain.
  The intensity of the pain of patients during a medical abortion will be quantified by a Visual Analogue Scale (VAS) at the time of the abortion and in the following 4 days.
  Groups: Group: Medical abortion with analgesic protocol
Other: Assessment of pain during voluntary termination of pregnancy by aspiration under local anesthesia following consideration of predictive factors of pain without an established analgesic protocol — Evaluation of the pain felt by women having an abortion by aspiration under local anesthesia.
  The intensity of the pain of patients during an abortion by aspiration under local anesthesia will be quantified by a Visual Analogue Scale (VAS) at the time of the abortion and in the following 4 days.Evaluation of the pain felt by women having an abortion by aspiration under local anesthesia.
  The intensity of the pain of patients during an abortion by aspiration under local anesthesia will be quantified by a Visual Analogue Scale (VAS) at the time of the abortion and in the following 4 days.
  Groups: Group: Abortion by aspiration under local anesthesia without analgesic protocol
Other: Assessment of pain during voluntary termination of pregnancy by aspiration under local anesthesia following consideration of predictive factors of pain with established analgesic protocol — Evaluation of the pain felt by women having an abortion by aspiration under local anesthesia following the application of an analgesic protocol indexed on the predictive factors of pain.
  The intensity of the pain of patients during an abortion by aspiration under local anesthesia will be quantified by a Visual Analogue Scale (VAS) at the time of the abortion and in the following 4 days.
  Groups: Group: Abortion by aspiration under local anesthesia with analgesic protocol

SUMMARY:
Two studies carried out in 2011 at the Center for Contraception and Voluntary Interruption of Pregnancy (CIVG) at the Louis-Mourier Hospital, evaluated the pain of patients undergoing an abortion, and looked for predictors of the pain felt during an abortion. medication or aspiration under local anesthesia.

These predictive factors of pain are today integrated into the interview during a request for abortion at the CIVG of Louis-Mourier.

This new study, on care data, prospective and monocentric conducted at the CIVG, of the Louis Mourier hospital, will make it possible to verify whether the knowledge of these predictive factors of pain has made it possible to improve the management of pain in women undergoing an abortion.

The main objective is to assess the pain felt by the patient during a medical abortion or by aspiration under local anesthesia, knowing the predictive factors of pain highlighted by two studies carried out in 2011.

The secondary objective is to highlight a significant difference in pain after application of an analgesic protocol indexed on predictive factors of pain.

The study will be carried out in two successive periods:

A first period of 4 months will consist in evaluating the pain felt by women having a medical abortion or by aspiration under local anesthesia.

A second period of 4 months will evaluate the pain felt by women undergoing medical or aspiration abortion under local anesthesia following the application of an analgesic protocol indexed on the predictive factors of pain.

The expected benefit of this study is the improvement of care and professional practices for better management of pain during outpatient abortion.

The abortion will take place in the usual way according to the chosen method. An information and non-objection note will be distributed to patients during the first consultation for an abortion.

Patients agreeing to participate in the study will answer the usual questions from the doctor or nurse.

A data collection sheet related to care will be integrated into the medical records. The CIVG doctors taking part in the study will report the data collected on this form.

The maximum pain felt during the abortion and in the following 4 days will be evaluated using an VAS according to usual practice.

DETAILED DESCRIPTION:
Procedure in two successive periods (Phase 1 and Phase 2) of 4 months each:

Phase 1: Evaluation of the pain felt by women undergoing medical or aspiration abortion under local anesthesia at the CIVG in Louis-Mourier.

Phase 2: Evaluation of the pain felt by women having a medical abortion or by aspiration under local anesthesia following the application of an analgesic protocol indexed on the predictive factors of pain at the CIVG of Louis-Mourier.

The progress of each of the phases is identical, only the management of the pain will be different.

During Phase 1, the analgesic choice will be left to the discretion of the doctor, as is already done at the CIVG of Louis Mourier.

During phase 2, analgesic management will be directed according to the presence of predictive factors of pain. The usual analgesics were integrated into an analgesic protocol indexed on the presence of predictive factors of pain.

ELIGIBILITY:
Inclusion Criteria:

* The population studied will concern all women over the age of 15 wishing to benefit from a medical abortion or by aspiration under local anesthesia.
* Understanding French orally, speaking it.
* Agreeing to participate in the study.

Exclusion Criteria:

* Unable to obtain information
* Not fluent in French
* Presenting complications (retention, clots) on the day of the abortion or after it.
* Aged under 15
* Refusing to participate in the study

Ages: 15 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Study on voluntary termination of pregnancy.
Study Population: All women over the age of 15, benefiting from a medical abortion or by aspiration under local anesthesia.
Sampling Method: Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the pain felt by the patient during a medical abortion or by aspiration under LA, knowing the predictive factors of pain highlighted by two studies carried out in 2011. | From the abortion to the follow-up visit two to four weeks after the abortion
  Pain VAS 0-100 mm (100 = worst pain)

SECONDARY OUTCOMES:
Highlight a significant difference in pain after application of an analgesic protocol indexed on predictive factors of pain. | From the abortion to the follow-up visit two to four weeks after the abortion
  Pain VAS 0-100 mm (100 = worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Soulat, docteur, Study Director — CIVG hôpital Louis Mourier
Locations (1):
- Centre d'Interruption Volontaire de Grossesse et de Contraception de l'Hôpital Louis Mourier, Colombes, France

IPD SHARING:
Plan to Share IPD: No